CLINICAL TRIAL: NCT05369520
Title: Non-invasive Spinal Cord Stimulation for Recovery of Autonomic Function After Spinal Cord Injury: Moving From Mechanisms to Clinical Practice
Brief Title: Non-invasive Spinal Cord Stimulation for Recovery of Autonomic Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrei Krassioukov, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H22-00365; CDMRP-SC210078 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2022-03-21; First posted 2022-05-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Autonomic Dysfunction; Sexual Dysfunction; Neurogenic Bladder Dysfunction; Neurogenic Bowel Dysfunction; Autonomic Dysreflexia; Orthostatic Hypotension
Keywords: Neurostimulation; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Primary Dysautonomias; Sexual Dysfunction, Physiological; Autonomic Dysreflexia; Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: Using a randomized counter-balanced approach, individuals will be allocated in two distinct pathways; the participants in Groups 1 (thoracic stimulation) and Group 2 (lumbosacral stimulation) will receive 8 weeks of TCSCS (3 times/week) at either mid/low thoracic or lumbosacral spinal cord levels respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Group 1 - Thoracic stimulation (Experimental): Participants will receive 8 weeks TCSCS at the mid/low thoracic spinal cord levels.
  Interventions: Device: TESCoN or SCONE device - Thoracic stimulation
- Group 2- Lumbosacral stimulation (Experimental): Participants will receive 8 weeks TCSCS at the lumbosacral spinal cord levels.
  Interventions: Device: TESCoN or SCONE device - Lumbosacral stimulation

INTERVENTIONS:
Device: TESCoN or SCONE device - Thoracic stimulation — TCSCS will be delivered using a non-invasive central nervous system stimulator (TESCoN or SCONE, SpineX Inc., CA, USA). The stimulation site will be over the thoracic spinal cord.
  Arms: Group 1 - Thoracic stimulation
Device: TESCoN or SCONE device - Lumbosacral stimulation — TCSCS will be delivered using a non-invasive central nervous system stimulator (TESCoN or SCONE, SpineX Inc., CA, USA). The stimulation site will be over the lumbosacral spinal cord.
  Arms: Group 2- Lumbosacral stimulation

SUMMARY:
This study is a pilot clinical trial to explore the efficacy of transcutaneous spinal cord stimulation (TCSCS) (proof-of-concept) in mitigating crucial autonomic dysfunctions that impact the health-related quality of life of individuals with spinal cord injury (SCI).

DETAILED DESCRIPTION:
This is a pilot clinical trial to explore the efficacy of TCSCS (proof-of-concept) in mitigating crucial autonomic dysfunctions that impact the health-related quality of life of individuals with SCI. A total of 30 eligible participants will be recruited and attend forty-two visits. All experiments will be performed at ICORD (Primary site) and the Brenda and David McLean Integrated Spine Clinic (SCI clinic), with the exception of anorectal manometry testing conducted at the Gastroenterology Clinic, St Paul's Hospital (GI clinic).

Following completion of screening and signing informed consent forms (visit 1), participants will undergo spatiotemporal mapping of spinal cord segments known to be involved in blood pressure, lower urinary tract and bowel control (visit 2). Following mapping, all individuals will undergo baseline functional assessments with and without TCSCS during 5 visits (visits 3-7), over a period of 4 weeks. To minimize the order effect, the functional assessments will be performed in a randomized order. Following baseline assessments, using a randomized counter-balanced approach, individuals will be allocated in two distinct pathways; the participants in Groups 1 and 2 will receive 8 weeks of TCSCS (3 times/week) at either mid/low thoracic or lumbosacral spinal cord levels respectively (visits 8- 31). Following long-term TCSCS, participants will undergo functional assessments during 5 visits (visits 32- 36) over a period of 4 weeks. In order to evaluate the persistent effects of TCSCS, all assessments will be repeated 8 weeks after cessation of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Resident of British Columbia, Canada with active provincial medical services plan.
2. Male or female, 19-60 years of age.
3. Chronic traumatic SCI (non-progressive, with complete motor paralysis) at or above the T6 spinal segment.
4. >1-year post injury, at least 6 months from any spinal surgery.
5. American Spinal Injury Association Impairment Scale (AIS) A, B.
6. Stable management of spinal cord related clinical issues (i.e., spasticity management).
7. Experience bladder, or bowel, or sexual dysfunction.
8. No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing.
9. For women of childbearing potential, not intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

   1. A confirmed negative pregnancy test prior to the baseline visit. During the trial, all women of childbearing potential will undergo urine pregnancy tests at their monthly clinic visits as outlined in the schedule of events.
   2. Use adequate contraception, or complete abstinence from sexual activities, during the period of the trial and for at least 28 days after completion of treatment.
   3. If using combined hormonal contraception, a stable regimen during the period of the trial and for at least 28 days after completion of treatment.
10. For sexually active males with female partners of childbearing potential, use adequate contraception, or complete abstinence from sexual activities, during the period of the trial and for at least 28 days after completion of treatment.
11. Must provide informed consent.
12. Willing and able to comply with all clinic visits and study-related procedures.
13. Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).

Exclusion Criteria:

1. Ventilator dependent.
2. Signs of lower motor neuron damage (i.e. concomitant conus medullaris/cauda equina injury).
3. Severe anemia or hypovolemia as measured by hematocrit via blood test in the last six months.
4. History of cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
5. History of seizures/epilepsy or recurring headaches.
6. Clinically significant, unmanaged, depression (to be screened) or ongoing drug abuse.
7. Intrathecal baclofen pump.
8. Oral baclofen dose greater than 60mg.
9. Individuals that have received intradetrusor or intrasphincter onabotulinumtoxinA injections within 6 months of baseline.
10. Any implanted metal (other than dental implants) in the skull or presence of pacemakers, stimulators, or medication pumps in the trunk.
11. Past electrode implantation surgery.
12. Member of the investigational team or his/her immediate family.
13. Presence of severe acute medical issue and use of any specific medication or treatment that, in the investigator's judgement, would adversely affect the participant's participation in the study.
14. Known allergies or sensitivities to both blue dye and beetroot powder.
15. Known or suspected gastrointestinal obstruction.
16. Persons with active inflammatory bowel disease or a history of bowel perforation.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Targeted TCSCS map modulate resting blood pressure (BP) | Week 1-2 (once)
  Using continuous beat-by beat BP monitoring via finger photoplethysmography during TCSCS, the researchers will identify the location and stimulation parameters to increase and decrease resting BP. Stimulation site will be either on the thoracic spinal cord (T7-T12) or the lumbosacral spinal cord (L1 - L3). Stimulation will be applied at various frequencies ranging between 1Hz and 90Hz. The outcome is an individualized TCSCS map (i.e. location and stimulation parameters) with change in systolic BP at rest during TCSCS.
Targeted TCSCS map to activate skeletal muscles and pelvic floor muscles | Week 1-2 (once)
  Using surface electromyography (EMG), the researchers will identify the motor threshold for skeletal muscles known to be involved in lower urinary tract, bowel and sexual control by delivering TCSCS at various spinal cord segments (T7 to conus medullaris). The outcome is an individualized TCSCS map (i.e. location and stimulation parameters) with pertinent motor thresholds for TCSCS-driven surface EMG.
Immediate change in BP during the head up tilt test (HUTT) | Week 3 - 6 (once)
  During HUTT, participants will be passively moved to approximately 60° upright stand position by the investigators using the tilt table. Using TCSCS to activate spinal sympathetic circuitry and mitigate low resting BP and orthostatic hypotension (OH), and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving OH triggered by HUTT.
Change in BP during the head up tilt test (HUTT) from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Using TCSCS and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of long-term TCSCS in improving OH triggered by HUTT.
Change in BP during the head up tilt test (HUTT) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Using TCSCS and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of long-term TCSCS in improving OH triggered by HUTT after cessation of therapy.
Immediate change in BP during digital anorectal stimulation (DARS) | Week 3 - 6 (once)
  DARS is a routine procedure to initiate a bowel routine. The participant will lay on their right side and DARS will be delivered via an index finger inserted into the rectum, applying gentle pressure for 30-60s. Utilizing TCSCS to inhibit nociceptive afferent and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving autonomic dysreflexia (AD) triggered by DARS.
Change in BP during digital anorectal stimulation (DARS) from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of long-term TCSCS in improving AD triggered by DARS.
Change in BP during digital anorectal stimulation (DARS) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of TCSCS in improving AD triggered by DARS after cessation of therapy.
Immediate change in rectal pressure measured by anorectal manometry (ARM) | Week 3 - 6 (once)
  ARM is well-established methodology that provides a direct assessment of anal sphincter pressure and anorectal coordination during simulated defecation. The test is performed by inserting a catheter, that contains a probe embedded with pressure sensors, through the anus and into the rectum. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing average max resting and squeeze pressure (mmHg).
Immediate change in high pressure anal canal zone measured by ARM | Week 3 - 6 (once)
  Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing length of high pressure anal canal zone (cm).
Immediate change in recto-anal inhibitory reflex measured by ARM | Week 3 - 6 (once)
  Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing recto-anal inhibitory reflex.
Immediate change in rectal sensation measured by ARM | Week 3 - 6 (once)
  Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing rectal sensation (mL).
Change in rectal pressure measured by ARM from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of long-term TCSCS in changing average max resting and squeeze pressure (mmHg).
Change in high pressure anal canal zone measured by ARM from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of long-term TCSCS in changing length of high pressure anal canal zone (cm).
Change in rectal sensation measured by ARM from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of long-term TCSCS in changing rectal sensation (mL).
Change in recto-anal inhibitory reflex measured by ARM from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of long-term TCSCS in changing recto-anal inhibitory reflex.
Change in rectal pressure measured by anorectal manometry (ARM) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of TCSCS in changing average max resting and squeeze pressure (mmHg).
Change in high pressure anal canal zone measured by anorectal manometry (ARM) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of TCSCS in changing length of high pressure anal canal zone (cm).
Change in recto-anal inhibitory reflex measured by anorectal manometry (ARM) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of TCSCS in changing recto-anal inhibitory reflex.
Change in rectal sensation measured by anorectal manometry (ARM) from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and ARM, researchers will test the safety and efficacy of TCSCS in changing rectal sensation (mL).
Immediate change in intravesical pressure at first sensation measured by urodynamic investigation (UDI) | Week 3 - 6 (once)
  Standard clinical procedures for UDI, including cystometry with water at 21°C and a filling rate of < 30 mL per minute through a 6F double lumen catheter with the participants in the supine position, provides a direct assessment of voiding and storage function. Abdominal pressure will be measured with a 10F intrarectal balloon catheter. Filling will be stopped when the participants report a sensation of fullness. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing intravesical pressure at first sensation (mmHg).
Immediate change in intravesical pressure at leakage point measured by UDI | Week 3 - 6 (once)
  Filling will be stopped at the moment of urine leakage. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing intravesical pressure at leakage point (mmHg).
Immediate change in intravesical pressure at maximal volume measured by UDI | Week 3 - 6 (once)
  Filling will be stopped at the moment of discomfort/per the request of patient. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly changing intravesical pressure at maximal volume (mmHg).
Change in intravesical pressure at first sensation measured by UDI from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of long-term TCSCS in changing intravesical pressure at first sensation (mmHg).
Change in intravesical pressure at leakage point measured by UDI from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of long-term TCSCS in changing intravesical pressure at leakage point (mmHg).
Change in intravesical pressure at maximal volume measured by UDI from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of long-term TCSCS in changing intravesical pressure at maximal volume (mmHg).
Change in intravesical pressure at first sensation measured by UDI from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of TCSCS in changing intravesical pressure at first sensation (mmHg).
Change in intravesical pressure at leakage point measured by UDI from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of TCSCS in changing intravesical pressure at leakage point (mmHg).
Change in intravesical pressure at maximal volume measured by UDI from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS and UDI, researchers will test the safety and efficacy of TCSCS in changing intravesical pressure at maximal volume (mmHg).
Immediate change in BP during penile or clitoral vibrostimulation | Week 3 - 6 (once)
  Genital vibration will be applied by an experienced physician using one or more handheld vibrators placed about the glans penis or the clitoral area with an amplitude of 1.0-3.5 mm and a frequency of 70-100 Hz. Utilizing TCSCS to inhibit nociceptive afferent and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of short-term TCS in reproducibly improving AD triggered by vibrostimulation.
Change in BP during penile or clitoral vibrostimulation from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of long-term TCSCS in improving AD triggered by vibrostimulation.
Change in BP during penile or clitoral vibrostimulation from baseline to 8 weeks after cessation of TCSCS | Week 27-30 (once)
  Utilizing TCSCS to inhibit nociceptive afferent and continuous beat-by beat BP monitoring via finger photoplethysmography, researchers will test the safety and efficacy of TCSCS in improving AD triggered by vibrostimulation.
Baseline assessment of colonic motility using the wireless motility capsule | Week 3 - 6 (once)
  The wireless motility capsule will be ingested and pass naturally through the GI tract, and data will be sent wirelessly to the data receiver. Researchers will use the collected data to assess baseline transit times.
Change in colonic motility using the wireless motility capsule from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Utilizing TCSCS and the wireless motility capsule, researchers will test the safety and efficacy of long-term TCSCS in improving transit times.
Change in colonic motility using the wireless motility capsule from baseline to 8 weeks after TCSCS cessation. | Week 27-30 (once)
  Utilizing TCSCS and the wireless motility capsule, researchers will test the safety and efficacy of TCSCS in improving transit times after cessation of therapy.

SECONDARY OUTCOMES:
Immediate change in cerebral blood flow (CBF) measured by trans-cranial doppler (TCD) during HUTT | Week 3 - 6 (once)
  TCD is a non-invasive ultrasound technique used to measure real-time CBF velocity. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving CBF during HUTT.
Change in CBF measured by TCD during HUTT from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Researchers will test the safety and efficacy of long-term TCSCS in improving CBF during HUTT.
Change in CBF measured by TCD during HUTT from baseline to 8 weeks after TCSCS cessation | Week 27-30 (once)
  Researchers will test the safety and efficacy of TCSCS in improving CBF during HUTT after cessation of therapy.
Immediate change in performance on the verbal fluency test (VFT) during HUTT | Week 3 - 6 (once)
  Phonetic/letter fluency, specifically total number of words, will be measured using the verbal fluency test (VFT). Researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving cognitive function during HUTT.
Change in performance on the VFT from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Researchers will test the safety and efficacy of long-term TCSCS in improving phonetic/letter fluency using the VFT.
Change in performance on the VFT from baseline to 8 weeks after TCSCS cessation | Week 27-30 (once)
  Researchers will test the safety and efficacy of TCSCS in improving phonetic/letter fluency after cessation of therapy.
Immediate change in performance on the Stroop Color and Word (SCW) test during HUTT | Week 3 - 6 (once)
  Ability to inhibit cognitive interference, specifically completion time, will be measured using the Stroop Color and Word (SCW) test. Researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving completion time of the SCW.
Change in performance on SCW from baseline to after completion of 8 weeks of TCSCS | Week 15-18 (once)
  Researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving completion time of the SCW.
Change in performance on SCW from baseline to 8 weeks after TCSCS cessation | Week 27-30 (once)
  Researchers will test the safety and efficacy of short-term TCSCS in reproducibly improving completion time of the SCW after cessation of therapy.

OTHER OUTCOMES:
Frequency of urinary incontinence will be measured using The Incontinence-Quality of Life (I-QoL) questionnaire. | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  Assessment of urinary incontinence will be performed to assess the impact of long term TCSCS on this measure. The scale is a 100 point scale where 0 is most severe incontinence.
Neurogenic bladder symptoms will be measured using the Neurogenic Bladder Symptom Score (NBSS). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  Assessment of neurogenic bladder symptoms will be performed to assess the impact of long term TCSCS on this measure. The score measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23), with higher scores representing worse symptoms.
Frequency of fecal incontinence will be measured using the modified Wexner Fecal Incontinence Score (WIS). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  Assessment of fecal incontinence will be performed to assess the impact of long term TCSCS on this measure. Scores can range from 0-20, with a higher score representing greater incontinence.
Neurogenic bowel symptoms will be measured using the Neurogenic Bowel Dysfunction (NBD) score. | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  Assessment of neurogenic bowel symptoms will be performed to assess the impact of long term TCSCS on this measure. Scores can range from 0-47, with a higher score representing more severe dysfunction.
Time Needed for Bowel Movement (TNFBM) will be measured by self-report. | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  Participants will be asked to record the time from 'suppository insertion' to 'when bowel evacuation is completed', during their regular bowel movement at home.
Participant's sexual function and satisfaction with their overall sexual life will be measured using the International Index of Erectile Function (IIEF-15). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  This measure of sexual function will be used to assess whether sexual function is impacted by TCSCS. Scores can range from 5-25, with higher scores representing greater function.
Participant's sexual function and satisfaction with their overall sexual life will be measured using the Female Sexual Function Index (FSFI). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  This measure of sexual function will be used to assess whether sexual function is impacted by TCSCS. Scores can range from 2-36, with higher scores representing greater function.
Participant's sexual function and satisfaction with their overall sexual life will be measured using a semi-structured qualitative interview. | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  This measure of sexual function will be used to assess whether sexual function is impacted by TCSCS.
Participant's sexually related personal distress will be measured using the Female Sexual Distress Scale (FSDS). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  The FSDS is a 13-item self-report measure of sexually related personal distress in women. The 13 items of the scale are scored on a 5-point Likert scale ranging from 0 (never) to 4 (always). The total score is calculated as the sum of the responses and ranges from 0 to 52, with higher scores indicating a greater level of distress. A score of ≥11 serves as a cut-off value for diagnosing women with sexual distress.
Participant's sensations associated with orgasm will be measured using the Orgasm Rating Scale (ORS). | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  The ORS is a 28 item self-report measure of phenomenological sensations associated with orgasm in men and women. Items are scored from 0 (not at all) 5 (extremely), with total scores ranging from 0 to 140, and higher scores indicating better function.
Participant's quality of life will be measured using the Short Form Health Survey (SF-36) | Week 3 - 6 (once), Week 15-18 (once), week 27-30 (once)
  The SF-36 consists of 8 domains pertaining to the respondents' experiences in the last 4 weeks. Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD, PhD, FRCPC, Principal Investigator — The University of British Columbia, International Collaboration on Repair Discoveries (ICORD)
Locations (2):
- Canada (2):
  - Blusson Spinal Cord Centre, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
The research team plans to deposit final de-identified research data at a community-based repository for SCI research, such as Open Data Commons for SCI (https://odc-sci.org//). Research resources, including but not limited to, established stimulation parameter and recording equipment, will also be made available through material transfer agreement upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available upon full-text print publication in a peer-reviewed journal, for a duration of at least 10 years.
Access Criteria: Online access or e-mail request to the corresponding author from an established scientific investigator